CLINICAL TRIAL: NCT02395081
Title: Trial of Vitamin D Supplements to Raise Calcidiol Levels of Pregnant Women in Mongolia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Maternal and Child Health Research, Mongolia (Unknown); Zuun Kharaa Hospital (Other)
Responsible Party: Principal Investigator, Janet Rich-Edwards, Director of Developmental Epidemiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 14-0591-02
Record Dates: First submitted 2015-02-11; First posted 2015-03-20 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Pregnancy; Vitamin D Deficiency
Keywords: pregnancy; Mongolia; Vitamin D; preeclampsia
MeSH Terms: conditions — Vitamin D Deficiency; Pre-Eclampsia | interventions — Cholecalciferol; Prenatal Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 600 IU (Placebo Comparator): Women will receive prenatal vitamins containing 600 IU of Vitamin D.
  Interventions: Dietary Supplement: 600 IU Vitamin D3 in prenatal vitamin
- 2000 IU (Experimental): Women will receive prenatal vitamins containing 2000 IU of Vitamin D.
  Interventions: Dietary Supplement: 2000 IU Vitamin D3 in prenatal vitamin
- 4000 IU (Experimental): Women will receive prenatal vitamins containing 4000 IU of Vitamin D.
  Interventions: Dietary Supplement: 4000 IU Vitamin D3 in prenatal vitamin

INTERVENTIONS:
Dietary Supplement: 600 IU Vitamin D3 in prenatal vitamin — Women will receive 600 IU 25(OH)D in prenatal vitamin.
  Arms: 600 IU
Dietary Supplement: 2000 IU Vitamin D3 in prenatal vitamin — Women will receive 2000 IU 25(OH)D in prenatal vitamin.
  Arms: 2000 IU
Dietary Supplement: 4000 IU Vitamin D3 in prenatal vitamin — Women will receive 4000 IU 25(OH)D in prenatal vitamin.
  Arms: 4000 IU

SUMMARY:
A double-blind randomized, placebo-controlled trial comparing the impact of 600 IU, 2000 IU, or 4000 IU of Vitamin D3 on third trimester 25(OH)D levels and change from baseline. The Vitamin D will be integrated in a standard prenatal vitamin, which will be taken from 12-16 weeks' gestation and continue throughout pregnancy. Umbilical cord 25(OH)D levels will also be determined. The investigators will generate preliminary data regarding Vitamin D intake and hypertensive disorders, blood pressure, and arterial function measured by tonography. The investigators will independently test blood pressure and proteinuria to identify preeclampsia cases.

DETAILED DESCRIPTION:
Vitamin D deficiency (serum 25(OH)D levels <20 ng/ml or 50 nmol/l) is widespread among Mongolians and is nearly universal during the winter months. The investigators have conducted a series of studies which have shown nearly universal Vitamin D deficiency in the winter months.

Observational studies in the U.S. have linked low 25(OH)D levels in women to a higher risk of preeclampsia. Mongolians also report levels of preeclampsia that are 3 times higher than those in the U.S (official reports cite 15%, though this may include gestational hypertension).

Given the widespread Vitamin D deficiency in Mongolian women, the high prevalence of hypertensive pregnancy in Mongolia, and the observational studies linking low 25(OH)D levels with preeclampsia risk, the investigators are conducting a pilot Vitamin D dosing trial to:

* Determine what level of Vitamin D supplementation is needed to secure 25(OH)D levels of at least 20 ng/ml in pregnant Mongolian women
* Generate preliminary data in support of a funding application for a larger trial of Vitamin D supplements to prevent preeclampsia in Mongolia

A double-blind randomized, placebo-controlled trial comparing the impact of 600 IU, 2000 IU, or 4000 IU of Vitamin D3 on third trimester 25(OH)D levels and change from baseline. The Vitamin D will be integrated in a standard prenatal vitamin, which will be taken from 12-16 weeks' gestation and continue throughout pregnancy. Umbilical cord 25(OH)D levels will also be determined. The investigators will generate preliminary data regarding Vitamin D intake and hypertensive disorders, blood pressure, and arterial function measured by tonography. The investigators will independently test blood pressure and proteinuria to identify preeclampsia cases.

The investigators will enroll 360 women who plan to receive their prenatal care and deliver at Zuun Kharaa Hospital in the Selenge province in northern Mongolia. Enrollment will be stratified by season. 120 women will be randomized to each of the three doses of vitamin D (600, 2000, 4000 IU) included in a standard prenatal vitamin.

Calcemia will be monitored two months after randomization and weeks 36-40 of pregnancy. Adverse events of pregnancy will be reported to the Data Safety and Monitoring Board (DSMB) and Institutional Review Board (IRB) per protocol.

Data will be gathered by a Mongolian study coordinator and local clinicians. A DSMB comprised of a U.S. and Mongolian clinicians and statisticians will monitor study data for safety.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* 12-16 weeks pregnant
* Receiving prenatal care at Zuun Kharaa Hospital and planning to deliver at Zuun Kharaa Hospital
* Willing not to take any additional vitamin D supplements, other than the study dispensed pills

Exclusion Criteria:

* Existing known seizure disorder, renal failure, parathyroid disease, thyroid disease, sarcoidosis, cancer, or tuberculosis. (Tuberculosis is routinely screened in pregnancy)
* History of kidney stones
* Known sensitivity to multivitamin preparations
* Taking vitamin D supplements containing >600 IU/day.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rich-Edwards, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Zuun Kharaa Hospital, Selenge, Selenge Province, Mongolia

REFERENCES:
- [Derived] Enkhmaa D, Tanz L, Ganmaa D, Enkhtur S, Oyun-Erdene B, Stuart J, Chen G, Carr A, Seely EW, Fitzmaurice G, Buyandelger Y, Sarantsetseg B, Gantsetseg G, Rich-Edwards J. Randomized trial of three doses of vitamin D to reduce deficiency in pregnant Mongolian women. EBioMedicine. 2019 Jan;39:510-519. doi: 10.1016/j.ebiom.2018.11.060. Epub 2018 Dec 11. PMID 30552064

RESULTS

PARTICIPANT FLOW:
Groups:
- 600 IU: Women will receive prenatal vitamins containing 600 IU of Vitamin D.
  Dietary supplement: 600 IU Vitamin D3 in prenatal vitamin
- 2000 IU: Women will receive prenatal vitamins containing 2000 IU of Vitamin D.
  Dietary supplement: 2000 IU Vitamin D in prenatal vitamin
- 4000 IU: Women will receive prenatal vitamins containing 4000 IU of Vitamin D.
  Dietary supplement: 4000 IU Vitamin D3 in prenatal vitamin
Period: Overall Study
Arm/Group | 600 IU | 2000 IU | 4000 IU
Started | 119 | 121 | 120
Completed | 112 | 116 | 116
Not Completed | 7 | 5 | 4
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Moved where blood couldn't be collected | 4 | 1 | 3
Not completed — Fetal Loss | 2 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 600 IU | 2000 IU | 4000 IU | Total
Number analyzed (Participants) | 119 | 121 | 120 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 119 | 121 | 120 | 360
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 121 | 120 | 360
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Serum 25(OH)D Concentration
Description: Circulating vitamin D at the end of the study as measured by VIDAS® enzyme linked fluorescent assay (ELFA)
Time Frame: 36 weeks gestation or delivery, if delivery occurred before 36 weeks
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 116 | 116
nmol/l | 46 (21) | 70 (23) | 81 (29)

2. Secondary Outcome: The Number of Participants With Preeclampsia
Description: Preeclampsia as measured by new onset hypertension after 20 weeks gestation and proteinuria.
Time Frame: After 20 weeks gestation
Population: Women delivering after 20 weeks in study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 116 | 117
Participants | 1 | 0 | 0

3. Secondary Outcome: Average Monthly Blood Pressure
Description: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) were measured in mm Hg at each antenatal care visit by the Study Coordinator, using the Omron- Elite 7300 (Omron Healthcare, Bannockburn, Illinois, USA) automated blood pressure monitor. Three blood pressure readings were taken after at least five minutes seated rest. For the analysis of mean blood pressures at each antenatal visit, the three readings were averaged for each participant.
Time Frame: During pregnancy
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 119 | 121 | 120
mmHg
  SBP wk 16-20 | 104.5 (9.2) | 104.5 (8.7) | 105.5 (9.7)
  SBP wk 20-24 | 105.1 (9.0) | 103.6 (8.2) | 105.4 (8.9)
  SBP wk 24-28 | 104.9 (9.1) | 103.3 (8.1) | 104.0 (9.3)
  SBP wk 28-32 | 104.5 (8.7) | 103.9 (9.7) | 105.4 (9.3)
  SBP wk 36-40 | 110.8 (10.1) | 110.6 (9.5) | 111.1 (11.0)
  DBP wk 16-20 | 63.8 (8.7) | 63.7 (8.7) | 65.2 (9.0)
  DBP wk 20-24 | 63.2 (9.0) | 63.1 (8.6) | 63.8 (9.6)
  DBP wk 24-28 | 64.2 (9.8) | 62.6 (9.4) | 63.5 (9.6)
  DBP wk 28-32 | 64.4 (8.7) | 63.6 (9.2) | 65.1 (9.2)
  DBP wk 32-36 | 67.2 (8.8) | 66.5 (9.4) | 67.1 (9.5)
  DBP wk 36-40 | 70.4 (9.7) | 71.0 (10.2) | 71.7 (10.6)
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.70, ANOVA — SBP wk 16-20

4. Secondary Outcome: Arterial Tonometry
Description: Investigators will assess Augmentation Index (AIx) and Pulse Wave Velocity (PWV) by study arm, as measured by AtCor Medical SphygmoCor device. THIS TONOMETER FAILED AND COULD NOT BE REPAIRED, SO WE ARE NOT PRESENTING THESE DATA AS OUTCOMES.
Time Frame: 36 weeks gestation
Reporting Status: Not Posted

5. Secondary Outcome: Number of Patients With Preterm Delivery as Measured by Clinical Diagnosis
Description: Gestational age was determined clinically by last menstrual period and by routine first trimester ultrasound which was universal; where these differed by more than 10 days, the ultrasound date was used. Gestational age at delivery was recorded by clinicians and rounded to the nearest week. Preterm delivery was defined as delivery before the 37th week of gestation.
Time Frame: During pregnancy
Population: Women delivering after 20 weeks at study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 116 | 117
Participants | 9 | 8 | 5
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.49, Chi-squared

6. Secondary Outcome: Casarean Section as Measured by Medical Record Abstraction
Description: Cesarean section was abstracted from the labor and delivery chart.
Time Frame: Delivery
Population: Women who delivered after 20 weeks at study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 116 | 117
Participants | 22 | 27 | 26
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.79, Chi-squared

7. Secondary Outcome: Assisted Vaginal Delivery as Measured by Medical Record Abstraction
Description: Assisted vaginal delivery with forceps delivery was abstracted from the labor and delivery chart.
Time Frame: Delivery
Population: Women who delivered after 20 weeks at the study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 116 | 117
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Small for Gestational Age (SGA) Neonates as Measured by Medical Record Abstraction
Description: SGA defined by the lowest 10th percentiles of sex-specific birthweight for gestational age charts of the INTERGROWTH-21st study
Time Frame: Delivery
Population: Singleton deliveries at study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 109 | 115 | 114
Participants | 1 | 2 | 2
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.83, Chi-squared

9. Secondary Outcome: Number of Large for Gestational Age (LGA) Neonates as Measured by Medical Record Abstraction
Description: LGA defined by the highest 10th percentiles of sex-specific birthweight for gestational age charts of the INTERGROWTH-21st study
Time Frame: Delivery
Population: Singleton deliveries after 20 weeks at study hospital
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 109 | 115 | 114
Participants | 25 | 26 | 33
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.39, Chi-squared

10. Secondary Outcome: Mean Calcemia as Measured by Serum Calcium Test (2mo)
Description: Measured on a semi-automated photometer (Humalyzer 3500, Human Diagnostics, Magdeburg, Germany)
Time Frame: 2 months after randomization
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 116 | 118 | 119
mmol/L | 2.2 (0.2) | 2.2 (0.2) | 2.2 (0.2)
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.24, ANOVA

11. Secondary Outcome: Number of Patients With Proteinuria as Measured by Urine Dipstick
Description: Proteinuria at last antenatal visit (usually 36-40 weeks' gestation), measured by 1+ Standard Diagnostics UroColor 10 10 (Kyonggi-do, South Korea) reagent strips
Time Frame: 36-40 weeks gestation/delivery
Population: Women who attended a last clinical visit after 36 weeks and gave a urine sample
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 92 | 93 | 87
Participants | 2 | 2 | 0
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.39, Chi-squared

12. Secondary Outcome: Number of Patients With Hypertensive Disorders of Pregnancy as Measured by Clinical Diagnosis
Description: In Mongolia, clinician-diagnosed preeclampsia may include a blood pressure increases >30 mm Hg above early pregnancy, with or without documented hypertension, proteinuria, or symptoms such as headache and edema
Time Frame: During pregnancy
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 119 | 121 | 120
Participants | 4 | 3 | 3
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.89, Chi-squared

13. Secondary Outcome: Number of Patients With Bacterial Vaginosis as Measured by Potassium Hydroxide (KOH) Wet Mount
Description: Bacterial vaginosis was routinely screened by potassium hydroxide wet mount at the first antenatal visit, at 28 weeks' and 32 weeks' gestation. It was also diagnosed by whiff test. We included both wet mount and whiff test positive in the bacterial vaginosis endpoint
Time Frame: During pregnancy
Population: Women seen for antenatal care during the trial
Measure: Count of Participants; unit: Participants
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 119 | 121 | 120
Participants | 17 | 19 | 18
Statistical Analysis 1: Comparison: 600 IU vs 2000 IU vs 4000 IU; Test type: Superiority; p = 0.95, Chi-squared

14. Secondary Outcome: Mean Calcemia as Measured by Serum Calcium Test (36-40 Weeks)
Description: Measured on a semi-automated photometer (Humalyzer 3500, Human Diagnostics, Magdeburg, Germany)
Time Frame: 36-40 weeks of pregnancy/delivery
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 600 IU | 2000 IU | 4000 IU
Number analyzed (Participants) | 112 | 113 | 113
mmol/L | 2.3 (0.2) | 2.3 (0.2) | 2.3 (0.2)

ADVERSE EVENTS:
Time Frame: From study enrollment (12-16 weeks gestation) to delivery
Description: Adverse events were reported by clinicians or by participants and recorded on standard forms reviewed by the study investigators and the Data Safety and Monitoring Board (DSMB). Antenatal care records were abstracted onto a standardized study form to record adverse events. The delivering clinician completed a checklist to record details and any adverse events of labor and delivery. The DSMB met every six months during the study to monitor study progress and safety.
Arm/Group | 600 IU | 2000 IU | 4000 IU
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/121 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/121 | 0/120
Other Adverse Events (participants affected / at risk) | 0/119 | 0/121 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes